CLINICAL TRIAL: NCT07030764
Title: Comparison of Arthrogenic Muscle Inhibition (AMI) After ACL Reconstruction in Patients With Conventional Rehabilitation or Conventional Rehabilitation Combined With Digital Therapy
Acronym: AMITHENUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-A00730-49
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation (Other): Conventional rehabilitation includes 40 physiotherapy sessions
  Interventions: Behavioral: Physiotherapy
- Aaugmented rehabilitation (Experimental): Augmented rehabilitation combines conventional rehabilitation (40 physiotherapy sessions) with the use of DOCT'UP® digital therapy.
  Interventions: Device: DOCT'UP

INTERVENTIONS:
Device: DOCT'UP — In addition to conventional physiotherapy sessions, DOCT'UP® is a mobile application which offers support programmes for patients following ACL reconstruction. This is digital therapy based on homebased physical exercises to be performed by patient.
  Arms: Aaugmented rehabilitation
Behavioral: Physiotherapy — Physiotherapy includes sessions performed at physiotherapist office under physiotherapist overview
  Arms: Conventional rehabilitation

SUMMARY:
Traumatic injury to the knee joint, such as rupture of the anterior cruciate ligament (ACL), can compromise the voluntary activation capacity of the quadriceps despite the anatomical integrity of the nerve and muscle structures responsible for contraction. This phenomenon is commonly known as 'arthrogenic muscle inhibition' (AMI).

AMI is a major limiting factor in recovery and rehabilitation after ACL rupture, and a potential cause of functional disability if left undiagnosed and untreated.

Traditional rehabilitation protocols for ACL reconstruction do not adequately address the underlying neuromuscular deficits caused by AMI, leading to sub-optimal recovery and prolonged rehabilitation. Furthermore, patient adherence to these protocols, outside of supervised settings, is variable and often poor, which can further delay recovery

Recent advances in digital health technologies offer new ways of improving rehabilitation outcomes. Numerous studies highlight the effectiveness of digital therapies in the form of mobile applications in improving patient engagement and compliance with rehabilitation protocols. In addition, evidence suggests that the integration of these technologies enables faster recovery of muscle function, reduces pain levels, may reduce complications such as Cyclops syndrome and improves overall patient satisfaction with rehabilitation.

Healing has developed a digital therapy called DOCT'UP® which, in addition to physiotherapy sessions, offers support programmes for patients following ACL reconstruction. These programmes include self-education exercises to be carried out at home, some of which specifically target the AMI phenomenon. DOCT'UP® digital therapy has already been used in rehabilitation after ACL reconstruction, with results at 3 weeks on quadriceps activation and post-operative pain, as well as at 1 year on Cyclops syndrome.

Given the limitations of current rehabilitation practices in the context of AMI and the potential of the DOCT'UP® application, there is a clear need to scientifically assess whether the DOCT'UP® application can effectively improve the results of rehabilitation on AMI after ACL reconstruction. This is why the sponsor wishes to set up this Clinical Investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years
* Patient with a scheduled primary ACL reconstruction
* Patient with a smartphone and able to use a mobile application on a smartphone
* Patient affiliated to or benefiting from a social security scheme
* French-speaking patient who has signed an informed consent form

Exclusion Criteria:

* Patients with residual AMI
* Patient with previous ipsi or contralateral knee surgery
* Patient with a multi-ligament injury
* Patient with contraindications to physical exercise: severe cardiovascular disease or uncontrolled metabolic disease
* Patients with cognitive problems
* Patient without internet access
* Patient taking part in another study
* Pregnant or breast-feeding women
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
AMI rate | 3 weeks
  The rate of patients with an AMI will be defined as a percentage of patients with AMI according to the Sonnery-Cottet classification (Sonnery-Cottet et al, 2022).
Physiotherapy adherence | 6 months
  Physiotherapy adherence will include number of physiotherapy sessions per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France, France

IPD SHARING:
Plan to Share IPD: No